CLINICAL TRIAL: NCT00158535
Title: Liver Transplantation in Patients With Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) Coinfection ANRS HC08 Thevic
Brief Title: Liver Transplantation in Patients With Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV) Coinfection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS HC08 THEVIC
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections; Hepatitis C
Keywords: Liver Transplantation; Hepatitis C; HIV Infections
MeSH Terms: conditions — HIV Infections; Hepatitis C | interventions — Liver Transplantation

INTERVENTIONS:
Procedure: liver transplantation

SUMMARY:
To show the feasibility of liver transplantation in HCV-HIV coinfected patients. To study the two-year survival after transplantation, the interaction between HCV and HIV after transplantation, the influence of HIV on HCV recurrence after transplantation, the interaction between immunosuppressive and antiretroviral drugs in particular anti-proteases, immunological follow-up and quality of life of these patients

DETAILED DESCRIPTION:
Until recently, HIV infection was considered as a contraindication for liver transplantation. A dramatic improvement in survival of HIV patients have been observed since the advent of new antiviral treatments against HIV including antiproteases. However an important proportion of patients with HCV-HIV coinfection are suffering from life-threatening liver disease due to HCV infection. Liver transplantation may be considered in this particular group of patients.

The ideal timing for the indication of liver transplantation during HIV disease and during the course of HCV liver disease needs to be defined. Liver transplantation in this particular group of patients raised several questions : a) the role of HIV infection on prevalence and severity of HCV recurrence after transplantation ; b) the role of liver transplantation and immunosuppression on HIV disease ; c) drug interactions between immunosuppressive agents and antiproteases ; d) immunological follow-up and quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Coinfection HIV-HVC
* Indication of liver transplantation for severe hepatopathy with life threatening:repetitive ascitis or infection of ascitis or icterus or decreased of prothrombin index under 50 percent or digestive haemorrhage by portal hypertension uncontrolled

Exclusion Criteria:

* Toxicomania
* Alcohol consumer (over 30g per day)
* AgHBs positive
* hepatocarcinoma over 5 cm or 3 nodules
* CD4 below 200/mm3
* Viral load below 400 cp
* HIV stade C

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2002-06

PRIMARY OUTCOMES:
Feasibility of liver transplantation in patients with HCV-HIV coinfection: survival at one and two years.

SECONDARY OUTCOMES:
Graft survival
Unexpected infections or neoplasia
Toxicity of antiretroviral and immunosuppressive treatments
Replicative kinetics of HIV and HVC after transplantation in blood and liver
Immune status of HIV and HVC
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Didier Samuel, MD, Principal Investigator — Hopital Paul Brousse Villejuif France; Bruno Fallisard, MD, Study Chair — Unité de Santé Publique, Hôpital Paul Brousse, Villejuif France
Locations (1):
- Centre hepato biliaire hopital paul Brousse, Villejuif, France